CLINICAL TRIAL: NCT00763269
Title: The Efficacy of a Toothpaste to Reduce Sensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-0208-TOT-SEN-PR
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2011-06

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Triclosan; Silicon Dioxide; Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): sensitive toothpaste
  Interventions: Drug: Triclosan, Silicon dioxide, fluoride
- B (Active Comparator): Triclosan control toothpaste
  Interventions: Drug: Triclosan, fluoride

INTERVENTIONS:
Drug: Triclosan, Silicon dioxide, fluoride — Brush twice daily
  Arms: A
Drug: Triclosan, fluoride — Brush twice daily
  Arms: B

SUMMARY:
Hypersensitivity

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages: 12 years or older.
* Availability for the eight-week duration of the study.
* Two sensitive teeth, which must be anterior to the molars, and demonstrate cervical erosion/abrasion or gingival recession.
* Qualifying response to Tactile stimuli (Yeaple Probe) as defined by a score between 10-50 grams of force.
* Qualifying response to the Air Blast stimuli as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both parameters assessed (Tactile or Air Blast) on at least two teeth to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for one month prior to entry into the study.
* Signed Informed Consent Form.

Exclusion Criteria:

* Gross oral pathology, chronic disease, or history of allergy to test products.
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with a mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Regular use of anticonvulsants, antihistamines, sedatives, tranquilizers, anti-inflammatory drugs, or analgesics.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past one month.
* Current participation in any other clinical study.
* Allergies to triclosan, or oral care products, personal care consumer products, or their ingredients.
* Medical condition which prohibits not eating/drinking for 4 hours.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Elias, DDS, Principal Investigator — Univ of Puerto Rico
Locations (1):
- Concordia Clinical Research, Cedar Knolls, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited by the PI at the clinical site
Pre-assignment Details: subjects were screened for medical and oral health criteria and then entered a 1 week washout before study treatment period.
Groups:
- A-Experimental Toothpatse: fluoride/triclosan/silica dioxide toothpaste (Sensitive teeth formula)
- B -Control Toothpaste: Fluoride/Triclosan control toothpaste
Period: Overall Study
Arm/Group | A-Experimental Toothpatse | B -Control Toothpaste
Started | 314 | 312
Completed | 302 | 299
Not Completed | 12 | 13
Not completed — Lost to Follow-up | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-Experimental Toothpatse | B -Control Toothpaste | Total
Number analyzed (Participants) | 314 | 312 | 626
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 2 | 9
  Between 18 and 65 years | 301 | 306 | 607
  >=65 years | 6 | 4 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 40.6 (13.4) | 41.4 (12.1) | 41 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 233 | 459
  Male | 88 | 79 | 167
Region of Enrollment [Number; unit: participants]
  United States | 314 | 312 | 626

OUTCOME MEASURES:

1. Primary Outcome: Hypersensitivity Tactile(Yeaple Probe)
Description: Measured with an electronic force sensing probe (Yeaple Probe): 10, 20, 30, 40, up to 50 grams of force are applied to hypersensitive tooth until pain elicited. Grams of force needed to elicit pain are recorded as hypersensitivity score for the tooth. For Tactile Hypersensitivity: The higher the score (the more grams of force needed to elicit a response of pain), the lower the hypersensitivity. Hypersensitivity scores on a per study subject basis are recorded as mean scores of two hypersensitive teeth
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A-Experimental Toothpatse | B -Control Toothpaste
Number analyzed (Participants) | 314 | 312
units on a scale | 19.81 (9.56) | 13.94 (6.42)
Statistical Analysis 1: Comparison: A-Experimental Toothpatse vs B -Control Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Hypersensitivity Tactile (Yeaple Probe)
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A-Experimental Toothpatse | B -Control Toothpaste
Number analyzed (Participants) | 314 | 312
Units on a scale | 31.90 (12.26) | 17.28 (8.86)
Statistical Analysis 1: Comparison: A-Experimental Toothpatse vs B -Control Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

3. Secondary Outcome: Air Blast Hypersensitivity (4 Week)
Description: Examiner rates the response to stimulation of hypersensitive teeth using a jet of air (constant stimulus on the basis of duration, pressure, temperature, distance from target). Response is rated based on the Schiff Cold Air Sensitivity Scale.This analog scale scores for the tooth is 0,1,2 or 3:"0"No subject response to stimulus"1"responds but will continue"2"responds and moves or requests discontinuation"3"Painful response to stimulus, discontinuation requested. The lower the score, the lower the hypersensitivity.Scores per study subject are recorded as mean scores of two hypersensitive teeth.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A-Experimental Toothpatse | B -Control Toothpaste
Number analyzed (Participants) | 314 | 312
units on a scale | 1.61 (0.62) | 2.18 (0.60)
Statistical Analysis 1: Comparison: A-Experimental Toothpatse vs B -Control Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

4. Secondary Outcome: Air Blast Hypersensitivity (8 Week)
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A-Experimental Toothpatse | B -Control Toothpaste
Number analyzed (Participants) | 314 | 312
units on a scale | 0.89 (0.69) | 1.80 (0.72)
Statistical Analysis 1: Comparison: A-Experimental Toothpatse vs B -Control Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | A-Experimental Toothpatse | B -Control Toothpaste
Serious Adverse Events (participants affected / at risk) | 0/314 | 0/312
Other Adverse Events (participants affected / at risk) | 3/314 | 4/312
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-Experimental Toothpatse (N=314) | B -Control Toothpaste (N=312)
Burning sensation of mucosa (General disorders) | 1 (1) | 1 (1) — subject reported burning sensation on tongue, cheeks and lips. subject discontinued during the 4 weeks visit.
Redness in Perioral area (possible allergic reaction) (General disorders) | 1 (1) | 0 (0) — subject observed redness in perioral area. visited dermatologist who diagnosed a possible allergic reaction and recommended to discontinue study toothpaste.
Physical Accidents w/ injuries (General disorders) | 1 (1) | 3 (4) — Several subjects reported accident. 1 had a workplace accident and was put on bedrest. 1 fell and broke wrist while walking.1 fell in backyard and broke a bone in left foot. adn 1 subject reported 2 events(a foot sprain and a broken left foot bone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less